CLINICAL TRIAL: NCT03102983
Title: Sensory-motor Interactions in the Perception of Vowels: a Study in Repetition - Suppression
Acronym: NEUROPHONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: GIPSA-LAB (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC16.026
Record Dates: First submitted 2017-03-23; First posted 2017-04-06 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: MRI, Functional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Volonteers (Experimental)
  Interventions: Other: MRI functional

INTERVENTIONS:
Other: MRI functional — vowels records and MRI session

SUMMARY:
The aim of our study is to show by fMRI the involvement of the motor system in the perception of speech, and more particularly how this implication is modulated by the degree of prototypicity of the stimuli.

DETAILED DESCRIPTION:
Each participant will undergo two visits:

Phase 1: The Gipsa-Lab Laboratory's Department of Speech and Cognition. This first visit will make it possible to make recordings of their vowel productions and to verify that the participants correspond to the criteria necessary for the study (passing the Edinburgh manual laterality test and auditory thresholds checked using a " An audiogram). It will also be an opportunity to provide them with the consent documents and the fact sheet, which will give them time to read it before the MRI exam. The duration of this first visit will be approximately 1 hour.

Phase 2: fMRI review in the 3Tesla MRI Unit at the Grenoble University Hospital Center. Participants will first undergo a medical examination in order to verify their absence of contraindication to the MRI examination. At the end of this medical examination, the consent of participation will be signed. The participants will then be able to carry out the MRI examination for a duration of about 1h15, then the behavioral judgment test of perceptual distance. The total duration of this second visit will be approximately 1h45.

ELIGIBILITY:
Inclusion Criteria:

* Medicall exam before MRI
* Pregnant Women
* Patients aged 18-45 years, Right-handed
* without neurologic and/or psychiatric troubles
* normal audition
* Audition normale
* French mother tongue
* Social security affiliation

Exclusion Criteria:

* protected person
* MRI contraindication
* claustrophobia
* respirtaory and cardiovascular pathology
* toxic substances taking

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the involvement of the speech motor system in the perception of vowels, using functional magnetic resonance imaging (fMRI). | One hour and forty five minutes
  fMRI measured

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre KRAINIK, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU Grenoble-Alpes, Grenoble, Isère, France

IPD SHARING:
Plan to Share IPD: No